CLINICAL TRIAL: NCT04652934
Title: Effectiveness of the Neural Mobilization on Upper Limb Functionality in Patients With Acquired Brain Injury: Randomized, Controlled, Multi-Centric, Single-Blind Clinical Trial
Brief Title: Effectiveness of the Neural Mobilization on Upper Limb Functionality in Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanesa Abuín (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor-Investigator, Vanesa Abuín, PhD students Thesis Director, Universidad Europea de Madrid
Organization: Universidad Europea de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUFA CEIC 20/154
Record Dates: First submitted 2020-10-08; First posted 2020-12-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hemiplegia and Hemiparesis; Acquired Brain Injury
Keywords: Acquired Brain Injury; Hemiplegia; Neural Mobilization; Upper limb
MeSH Terms: conditions — Hemiplegia; Paresis; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Upper Limb Neurodynamic Test (ULNT1) technique described by Butler will be performed on the affected limb. This technique consists of performing shoulder depression, 90º shoulder abduction, hand, wrist and forearm in a neutral position, external rotation of the shoulder and extension of the elbow. After positioning the limb in this position, wrist flexion-extension movements will be performed smoothly and rhythmically of 20 movements every minute, for 3 minutes, three times per session with 1 minute of rest between each series.
  Interventions: Other: Neurodynamic
- Mimic group (Sham Comparator): The protocol used by Beneciuk et al. Will be used. This intervention consists of imitating NM without stressing the nervous system. It will be carried out as follow: a neutral cervical position will be maintained (0º of cervical inclination), 45º of shoulder abduction without depression, 45º of external rotation of the shoulder combined with 45º of elbow flexion with the forearm in pronation. Afterwards, 10 wrist flexion-extension movements will be performed at a rate of 6 seconds per cycle (3 seconds of flexion and 3 seconds of extension). The resistance that you will feel will stabilize when you change motion. Once the 10 cycles of movements have been carried out, a wrist flexion will be maintained for 10 seconds.
  Interventions: Other: Mimic group

INTERVENTIONS:
Other: Neurodynamic — The Upper Limb Neurodynamic Test (ULNT1) technique described by Butler will be performed on the affected limb. This technique consists of performing shoulder depression, 90º shoulder abduction, hand, wrist and forearm in a neutral position, external rotation of the shoulder and extension of the elbow. After positioning the limb in this position, wrist flexion-extension movements will be performed smoothly and rhythmically of 20 movements every minute, for 3 minutes, three times per session with 1 minute of rest between each series.
  Arms: Intervention group
Other: Mimic group — The protocol used by Beneciuk et al. Will be used. This intervention consists of imitating NM without stressing the nervous system. It will be carried out as follow: a neutral cervical position will be maintained (0º of cervical inclination), 45º of shoulder abduction without depression, 45º of external rotation of the shoulder combined with 45º of elbow flexion with the forearm in pronation. Afterwards, 10 wrist flexion-extension movements will be performed at a rate of 6 seconds per cycle (3 seconds of flexion and 3 seconds of extension). The resistance that you will feel will stabilize when you change motion. Once the 10 cycles of movements have been carried out, a wrist flexion will be maintained for 10 seconds.
  Arms: Mimic group

SUMMARY:
The main objective:

To determine changes in physiological and structural properties of upper limb muscles with spasticity in patients with acquired brain injury after applying neural mobilization improving their functional performance, their participation in society and quality of life.

Hypothesis:

Peripheral nerve mobilizations performed with neurodynamic techniques in upper limb in patients with acquired brain injury, generate changes at structural and physiological level, favoring the performance of daily life activities and improving the quality of life.

DETAILED DESCRIPTION:
Randomized clinical trial with blinding of the subject, the evaluator and the person analyzing the data.

In the experimental group will be performed neural mobilitazion technique, while in the sham a technique to mimic neurodynamic.

The assessment will be made by a single evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acquired brain injury (hemiplegia-hemiparesis)
* Ages between 25 and 50 years

Exclusion Criteria:

* Unable to understand and respond to verbal instructions
* Absence of voluntary movement in the upper limb
* Take medicine for spasticity
* Botulinum toxin infiltration in the last 6 months

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in Manual Ability | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  Abilhand Scale; Score 0(worse outcome)-2(better outcome)
Changes in Muscle Spasticity | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  MAS (Modified Ashworth Scale) 0 (better outcome) - 4 (worse outcome)
Changes in Muscle Strength | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  Dynamometer
Changes in Nervous Conduction | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  Delsys Trigno Avanti (surface eMG for non-invasive assessment of muscles)
Changes in Upper Limb Pain Perception | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  EVA (Visual Analog Scale) 0 (worse outcome) - 10 (better outcome)
Changes in Upper Limb Pain to Pressure | Pre-intervention; Immediately after the intervention; Follow up (1 week after the intervention)
  Algometer

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa Abuín, Dr, Study Chair — Universidad Europea de Madrid; Leticia Martínez, Dr, Study Director — Universidad Europea de Madrid; Almudena Buesa, Dr, Study Chair — Universidad San Jorge de Zaragoza
Locations (1):
- Federico Salniccia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The World Health report 1996--fighting disease, fostering development. World Health Forum. 1997;18(1):1-8. PMID 9233055
- [Background] Synnot A, Chau M, Pitt V, O'Connor D, Gruen RL, Wasiak J, Clavisi O, Pattuwage L, Phillips K. Interventions for managing skeletal muscle spasticity following traumatic brain injury. Cochrane Database Syst Rev. 2017 Nov 22;11(11):CD008929. doi: 10.1002/14651858.CD008929.pub2. PMID 29165784
- [Background] Basson A, Olivier B, Ellis R, Coppieters M, Stewart A, Mudzi W. The Effectiveness of Neural Mobilization for Neuromusculoskeletal Conditions: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Sep;47(9):593-615. doi: 10.2519/jospt.2017.7117. Epub 2017 Jul 13. PMID 28704626
- [Background] Martins C, Pereira R, Fernandes I, Martins J, Lopes T, Ramos L, Pacheco J, Silva AG. Neural gliding and neural tensioning differently impact flexibility, heat and pressure pain thresholds in asymptomatic subjects: A randomized, parallel and double-blind study. Phys Ther Sport. 2019 Mar;36:101-109. doi: 10.1016/j.ptsp.2019.01.008. Epub 2019 Jan 23. PMID 30710858
- [Background] Beltran-Alacreu H, Jimenez-Sanz L, Fernandez Carnero J, La Touche R. Comparison of Hypoalgesic Effects of Neural Stretching vs Neural Gliding: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2015 Nov-Dec;38(9):644-652. doi: 10.1016/j.jmpt.2015.09.002. Epub 2015 Oct 23. PMID 26481666
- [Background] Almeida RS, Machado E, Yamato TP, Santos De Melo L, Nogueira LAC. Pragmatic neural tissue management improves short-term pain and disability in patients with sciatica: a single-arm clinical trial. J Man Manip Ther. 2019 Sep;27(4):208-214. doi: 10.1080/10669817.2019.1580420. Epub 2019 Feb 26. PMID 30935325
- [Background] Ayub A, Osama M, Ahmad S. Effects of active versus passive upper extremity neural mobilization combined with mechanical traction and joint mobilization in females with cervical radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(5):725-730. doi: 10.3233/BMR-170887. PMID 30664500
- [Background] Kim DG, Chung SH, Jung HB. The effects of neural mobilization on cervical radiculopathy patients' pain, disability, ROM, and deep flexor endurance. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):951-959. doi: 10.3233/BMR-140191. PMID 28453446
- [Background] Ferragut-Garcias A, Plaza-Manzano G, Rodriguez-Blanco C, Velasco-Roldan O, Pecos-Martin D, Oliva-Pascual-Vaca J, Llabres-Bennasar B, Oliva-Pascual-Vaca A. Effectiveness of a Treatment Involving Soft Tissue Techniques and/or Neural Mobilization Techniques in the Management of Tension-Type Headache: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Feb;98(2):211-219.e2. doi: 10.1016/j.apmr.2016.08.466. Epub 2016 Sep 10. PMID 27623523
- [Background] Sanz DR, Solano FU, Lopez DL, Corbalan IS, Morales CR, Lobo CC. Effectiveness of median nerve neural mobilization versus oral ibuprofen treatment in subjects who suffer from cervicobrachial pain: a randomized clinical trial. Arch Med Sci. 2018 Jun;14(4):871-879. doi: 10.5114/aoms.2017.70328. Epub 2017 Sep 26. PMID 30002707
- [Background] Rodriguez-Sanz D, Calvo-Lobo C, Unda-Solano F, Sanz-Corbalan I, Romero-Morales C, Lopez-Lopez D. Cervical Lateral Glide Neural Mobilization Is Effective in Treating Cervicobrachial Pain: A Randomized Waiting List Controlled Clinical Trial. Pain Med. 2017 Dec 1;18(12):2492-2503. doi: 10.1093/pm/pnx011. PMID 28340157
- [Background] Rodriguez-Sanz D, Lopez-Lopez D, Unda-Solano F, Romero-Morales C, Sanz-Corbalan I, Beltran-Alacreu H, Calvo-Lobo C. Effects of Median Nerve Neural Mobilization in Treating Cervicobrachial Pain: A Randomized Waiting List-Controlled Clinical Trial. Pain Pract. 2018 Apr;18(4):431-442. doi: 10.1111/papr.12614. Epub 2017 Nov 20. PMID 28734105
- [Background] Arumugam V, Selvam S, MacDermid JC. Radial nerve mobilization reduces lateral elbow pain and provides short-term relief in computer users. Open Orthop J. 2014 Oct 17;8:368-71. doi: 10.2174/1874325001408010368. eCollection 2014. PMID 25352930
- [Background] Lau YN, Ng J, Lee SY, Li LC, Kwan CM, Fan SM, Leung BPL, Lo CN. A brief report on the clinical trial on neural mobilization exercise for joint pain in patients with rheumatoid arthritis. Z Rheumatol. 2019 Jun;78(5):474-478. doi: 10.1007/s00393-018-0521-7. PMID 30112581
- [Background] Villafane JH, Cleland JA, Fernandez-de-Las-Penas C. The effectiveness of a manual therapy and exercise protocol in patients with thumb carpometacarpal osteoarthritis: a randomized controlled trial. J Orthop Sports Phys Ther. 2013 Apr;43(4):204-13. doi: 10.2519/jospt.2013.4524. Epub 2013 Mar 13. PMID 23485660
- [Background] Veras LS, Vale RG, Mello DB, Castro JA, Lima V, Trott A, Dantas EH. Electromyography function, disability degree, and pain in leprosy patients undergoing neural mobilization treatment. Rev Soc Bras Med Trop. 2012 Feb;45(1):83-8. doi: 10.1590/s0037-86822012000100016. PMID 22370834
- [Background] Casanova C, Lerma Lara S, Perez Ruiz M, Ruano Dominguez D, Santana Sosa E. Non-pharmacological treatment for neuropathic pain in children with cancer. Med Hypotheses. 2015 Dec;85(6):791-7. doi: 10.1016/j.mehy.2015.10.007. Epub 2016 Oct 17. PMID 26604028
- [Background] Santos FM, Silva JT, Rocha IRC, Martins DO, Chacur M. Non-pharmacological treatment affects neuropeptide expression in neuropathic pain model. Brain Res. 2018 May 15;1687:60-65. doi: 10.1016/j.brainres.2018.02.034. Epub 2018 Feb 26. PMID 29496478
- [Background] Zhu GC, Tsai KL, Chen YW, Hung CH. Neural Mobilization Attenuates Mechanical Allodynia and Decreases Proinflammatory Cytokine Concentrations in Rats With Painful Diabetic Neuropathy. Phys Ther. 2018 Apr 1;98(4):214-222. doi: 10.1093/ptj/pzx124. PMID 29309710
- [Background] Santos FM, Grecco LH, Pereira MG, Oliveira ME, Rocha PA, Silva JT, Martins DO, Miyabara EH, Chacur M. The neural mobilization technique modulates the expression of endogenous opioids in the periaqueductal gray and improves muscle strength and mobility in rats with neuropathic pain. Behav Brain Funct. 2014 May 13;10:19. doi: 10.1186/1744-9081-10-19. PMID 24884961
- [Background] Giardini AC, Dos Santos FM, da Silva JT, de Oliveira ME, Martins DO, Chacur M. Neural Mobilization Treatment Decreases Glial Cells and Brain-Derived Neurotrophic Factor Expression in the Central Nervous System in Rats with Neuropathic Pain Induced by CCI in Rats. Pain Res Manag. 2017;2017:7429761. doi: 10.1155/2017/7429761. Epub 2017 Mar 22. PMID 28420943
- [Background] Santos FM, Silva JT, Giardini AC, Rocha PA, Achermann AP, Alves AS, Britto LR, Chacur M. Neural mobilization reverses behavioral and cellular changes that characterize neuropathic pain in rats. Mol Pain. 2012 Jul 29;8:57. doi: 10.1186/1744-8069-8-57. PMID 22839415
- [Background] da Silva JT, Santos FM, Giardini AC, Martins Dde O, de Oliveira ME, Ciena AP, Gutierrez VP, Watanabe IS, Britto LR, Chacur M. Neural mobilization promotes nerve regeneration by nerve growth factor and myelin protein zero increased after sciatic nerve injury. Growth Factors. 2015 Feb;33(1):8-13. doi: 10.3109/08977194.2014.953630. Epub 2014 Dec 9. PMID 25489629
- [Background] Nunes MK, Fontenele Dos Santos G, Martins E Silva DC, Mota de Freitas AC, Henriques IF, Andrade PM, Machado Dde C, Teixeira S, Neves MO, Dias G, Silva-Junior F, Bastos VH. Acute effects of neural mobilization and infrared on the mechanics of the median nerve. J Phys Ther Sci. 2016 Jun;28(6):1720-3. doi: 10.1589/jpts.28.1720. Epub 2016 Jun 28. PMID 27390402
- [Background] Neal Hanney R, Ridehalgh C, Dawson A, Lewis D, Kenny D. The effects of neurodynamic straight leg raise treatment duration on range of hip flexion and protective muscle activity at P1. J Man Manip Ther. 2016 Feb;24(1):14-20. doi: 10.1179/2042618613Y.0000000049. PMID 27252578
- [Background] Sharma S, Balthillaya G, Rao R, Mani R. Short term effectiveness of neural sliders and neural tensioners as an adjunct to static stretching of hamstrings on knee extension angle in healthy individuals: A randomized controlled trial. Phys Ther Sport. 2016 Jan;17:30-7. doi: 10.1016/j.ptsp.2015.03.003. Epub 2015 Mar 17. PMID 26482098
- [Background] Beneciuk JM, Bishop MD, George SZ. Effects of upper extremity neural mobilization on thermal pain sensitivity: a sham-controlled study in asymptomatic participants. J Orthop Sports Phys Ther. 2009 Jun;39(6):428-38. doi: 10.2519/jospt.2009.2954. PMID 19487826
- [Background] Calvo-Lobo C, Unda-Solano F, Lopez-Lopez D, Sanz-Corbalan I, Romero-Morales C, Palomo-Lopez P, Seco-Calvo J, Rodriguez-Sanz D. Is pharmacologic treatment better than neural mobilization for cervicobrachial pain? A randomized clinical trial. Int J Med Sci. 2018 Mar 8;15(5):456-465. doi: 10.7150/ijms.23525. eCollection 2018. PMID 29559834
- [Background] Brown CL, Gilbert KK, Brismee JM, Sizer PS, Roger James C, Smith MP. The effects of neurodynamic mobilization on fluid dispersion within the tibial nerve at the ankle: an unembalmed cadaveric study. J Man Manip Ther. 2011 Feb;19(1):26-34. doi: 10.1179/2042618610Y.0000000003. PMID 22294851
- [Background] Gilbert KK, Roger James C, Apte G, Brown C, Sizer PS, Brismee JM, Smith MP. Effects of simulated neural mobilization on fluid movement in cadaveric peripheral nerve sections: implications for the treatment of neuropathic pain and dysfunction. J Man Manip Ther. 2015 Sep;23(4):219-25. doi: 10.1179/2042618614Y.0000000094. PMID 26917940
- [Background] Kim MK, Cha HG, Ji SG. The initial effects of an upper extremity neural mobilization technique on muscle fatigue and pressure pain threshold of healthy adults: a randomized control trial. J Phys Ther Sci. 2016 Mar;28(3):743-6. doi: 10.1589/jpts.28.743. Epub 2016 Mar 31. PMID 27134351
- [Background] Castilho J, Ferreira LAB, Pereira WM, Neto HP, Morelli JGDS, Brandalize D, Kerppers II, Oliveira CS. Analysis of electromyographic activity in spastic biceps brachii muscle following neural mobilization. J Bodyw Mov Ther. 2012 Jul;16(3):364-368. doi: 10.1016/j.jbmt.2011.12.003. Epub 2012 Jan 20. PMID 22703748
- [Background] Godoi J, Kerppers II, Rossi LP, Correa FI, Costa RV, Correa JC, Oliveira CS. Electromyographic analysis of biceps brachii muscle following neural mobilization in patients with stroke. Electromyogr Clin Neurophysiol. 2010 Jan-Feb;50(1):55-60. PMID 20349559
- [Background] Ferreira J, Bebiano A, Raro D, Martins J, Silva AG. Comparative Effects of Tensioning and Sliding Neural Mobilization on Static Postural Control and Lower Limb Hop Testing in Football Players. J Sport Rehabil. 2019 Nov 1;28(8):840-846. doi: 10.1123/jsr.2017-0374. PMID 30222495
- [Background] Penta M, Tesio L, Arnould C, Zancan A, Thonnard JL. The ABILHAND questionnaire as a measure of manual ability in chronic stroke patients: Rasch-based validation and relationship to upper limb impairment. Stroke. 2001 Jul;32(7):1627-34. doi: 10.1161/01.str.32.7.1627. PMID 11441211
- [Background] Chuang LL, Wu CY, Lin KC, Lur SY. Quantitative mechanical properties of the relaxed biceps and triceps brachii muscles in patients with subacute stroke: a reliability study of the myoton-3 myometer. Stroke Res Treat. 2012;2012:617694. doi: 10.1155/2012/617694. Epub 2012 Apr 30. PMID 22619740
- [Background] Li F, Wu Y, Li X. Test-retest reliability and inter-rater reliability of the Modified Tardieu Scale and the Modified Ashworth Scale in hemiplegic patients with stroke. Eur J Phys Rehabil Med. 2014 Feb;50(1):9-15. Epub 2013 Dec 5. PMID 24309501
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Brinkmann JR. Comparison of a hand-held and fixed dynamometer in measuring strength of patients with neuromuscular disease. J Orthop Sports Phys Ther. 1994 Feb;19(2):100-4. doi: 10.2519/jospt.1994.19.2.100. PMID 8148862
- [Background] Trampisch US, Franke J, Jedamzik N, Hinrichs T, Platen P. Optimal Jamar dynamometer handle position to assess maximal isometric hand grip strength in epidemiological studies. J Hand Surg Am. 2012 Nov;37(11):2368-73. doi: 10.1016/j.jhsa.2012.08.014. PMID 23101534
- [Background] Price CI, Curless RH, Rodgers H. Can stroke patients use visual analogue scales? Stroke. 1999 Jul;30(7):1357-61. doi: 10.1161/01.str.30.7.1357. PMID 10390307
- [Background] Benaim C, Froger J, Cazottes C, Gueben D, Porte M, Desnuelle C, Pelissier JY. Use of the Faces Pain Scale by left and right hemispheric stroke patients. Pain. 2007 Mar;128(1-2):52-8. doi: 10.1016/j.pain.2006.08.029. Epub 2006 Oct 5. PMID 17027154
- [Background] Pelfort X, Torres-Claramunt R, Sanchez-Soler JF, Hinarejos P, Leal-Blanquet J, Valverde D, Monllau JC. Pressure algometry is a useful tool to quantify pain in the medial part of the knee: an intra- and inter-reliability study in healthy subjects. Orthop Traumatol Surg Res. 2015 Sep;101(5):559-63. doi: 10.1016/j.otsr.2015.03.016. Epub 2015 May 27. PMID 26025162
- [Background] Kostek M, Polaski A, Kolber B, Ramsey A, Kranjec A, Szucs K. A Protocol of Manual Tests to Measure Sensation and Pain in Humans. J Vis Exp. 2016 Dec 19;(118):54130. doi: 10.3791/54130. PMID 28060280
- [Derived] Salniccia F, Castel-Sanchez M, Bermejo-Franco A, Buesa-Estellez A, Lopez-Ruiz J, Abuin-Porras V. Preparatory use of neurodynamics to enhance upper limb function in patients with acquired brain injury: a randomized controlled trial. Sci Rep. 2025 Nov 29;16(1):159. doi: 10.1038/s41598-025-29095-y. PMID 41318749
- See also: Las personas con Daño Cerebral Adquirido en España — https://fedace.org/index.php?&PHPSESSID=3j4ek0jllf4n07r3qvb140nki4&V_dir=MSC&V_mod=download&f=2016-9/26-16-4-11.admin.Informe_FEDACE_RPD_para_DDC-1.pdf